CLINICAL TRIAL: NCT03856190
Title: Effectiveness of Therapeutic Fasting and Specific Diet in Patients With Rheumatoid Arthritis: a Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Therapeutic Fasting and Specific Diet in Patients With Rheumatoid Arthritis
Acronym: NutriFast
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid pandemic, research halt, expiring funding
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Braunschweig Integrated Centre of Systems Biology (BRICS), Germany (Unknown); University of Luxembourg (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NutriFast
Record Dates: First submitted 2019-01-24; First posted 2019-02-27 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2021-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Fasting; Vegan; Plant based; Randomized Trial
MeSH Terms: conditions — Arthritis, Rheumatoid; Fasting | interventions — Diet, Plant-Based

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting and "best practice" nutrition (Active Comparator): Initial fasting followed by 11 weeks plant-based diet
  Interventions: Other: Fasting and plant-based nutrition
- Standard Nutrition Counselling (Active Comparator): 12 weeks standard antiinflammatory diet
  Interventions: Other: Standard Nutrition Counselling

INTERVENTIONS:
Other: Fasting and plant-based nutrition — The experimental intervention is divided into an initial part with periodic fasting for 7-10 days on an outpatient basis, which is followed by a build-up phase. This group part then receives a diet change with a specific normocaloric nutrition including the concept of time restricted eating (TRE, 16/8h) and according to the following criteria: 1) plant-based, 2) rich in prebiotics, 3) enriched with kitchen spices and kitchen herbs known for their anti-mycotic and anti-inflammatory potential.
  Arms: Fasting and "best practice" nutrition
Other: Standard Nutrition Counselling — The control group receives a diet considered to be fundamentally beneficial to health in the sense of the recommendations of the German Association for Nutrition (DGE), which contain a reduced intake of arachidonic acid and, as a result, modulate an anti-inflammatory effect.
  Arms: Standard Nutrition Counselling

SUMMARY:
The aim of this trial is an evaluation of the effectiveness of fasting and a subsequent diagnosis-specific diet change in patients with rheumatoid arthritis in respect to improving rheumatic symptoms and further to investigate possible mechanisms of this improvement.

DETAILED DESCRIPTION:
Rheumatoid arthritis is an inflammatory-destructive joint disease for which up to date etiopathogenetical causes are lacking. In recent years, numerous new therapeutic concepts have been developed in the form of targeted antibody therapies that can block various inflammatory mechanisms. Although better treatment successes in comparison with conventional therapies were achieved, patients respond to the new therapies in very different ways. As a result the optimal drug needs to be identified for each patient through individual treatment trials. So far, no healings have been achieved and the progression of the disease can be stopped only by permanent suppression of the inflammatory response. In addition to different immunological mechanisms and genetic predispositions, interactions with the microbiome of the intestine are increasingly being discussed in recent years. A dysbiotic intestinal flora, characterized by the loss of beneficial bacteria and a concomitant increase in potentially pathogenic microbes, is associated with chronic inflammatory syndromes.

Modified fasting (up to 500 kcal energy intake per day) for 7-10 days leads to an improvement of the symptoms in many patients with rheumatoid arthritis and is regularly used by the applicants for the treatment of rheumatoid arthritis. Several clinical studies have shown that therapeutic fasting produces anti-inflammatory effects. However, so far no standardized method for long-term stabilization of corresponding effects after resumption of nutrition has been established.

Recent transcriptome analyzes have not only revealed numerous new potential markers, but also increasingly allow conclusions to be drawn from these extensive datasets that suggest immunological relationships between specific genes. In preliminary studies within the framework of a project of the same study group, it was possible to identify inflammatory profiles of individual foods and to identify molecular markers of disease activity in rheumatoid arthritis whose diagnostic value has been tested and interpreted under the influence of fasting. These markers will now be clinically evaluated in this study in collaboration with both centers.

The hypothesis is that a combination of fasting and subsequent diagnosis-specific diet change will improve the rheumatic symptoms. In this context, it will also be analyzed, which meaning of the changes 1) of the metabolism and 2) of the microbiome, mediated by fasting and nutrition, belongs. This will be demonstrated by using already identified markers for genotypic traits, gene expression traits, characteristics of protein expression, protein activities, and antigen-specific immunological response patterns.

The present research project aims to combine the different aspects of a possible anti-rheumatic nutrition and to evaluate the nutritherapeutic concept in an RCT. We suggest that a part of the anti-inflammatory effects of fasting and best practice diets may be due to a change in the composition of the intestinal flora mediated. Thus this study contributes to the extended therapy of rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Rheumatoid arthritis
2. free of any serious medical condition that precludes safe participation in an exercise program, such as coronary artery disease, severe hypertension, peripheral vascular disease, stroke, congestive heart failure, chronic obstructive pulmonary disease, insulin-dependent diabetes, psychiatric disease, renal disease, liver disease, active cancer other than skin cancer, and anemia
3. Ability to understand the intervention concept and written consent to participate;
4. Willingness to accept randomization and undergo the testing and intervention procedures and deliver stool, blood and urine samples for testing
5. Age 18-70 years (inclusive)
6. drug therapy was not started in the last 8 weeks before screening

Exclusion Criteria:

1. Gout or septic arthritis
2. Psychiatric disease that interferes with the understanding and implementation of the intervention
3. Pregnancy or breast feeding
4. In the case of pronounced anemia (Hb <10 mg / dl) no inclusion in the examination or no additional blood sampling is carried out
5. Underweight (BMI <18,5) or weight loss of >3kg/5kg in the last/last 3 month(s)
6. Eating disorder (such as bulimia, anorexia nervosa) in the last 5 years
7. Current vegan nutrition
8. Non-existence of email address or internet access

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Health Assessement Questionnaire (HAQ) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
  Change from Baseline in the HAQ after 12 weeks, range from 0 to 3 while higher values meaning a higher grade of disability

SECONDARY OUTCOMES:
Disease Activity Score 28 (DAS-28-CRP) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
  Change from Baseline in the DAS-28-CRP, range from 2.0 to 10.0 while higher values meaning a higher disease activity and below of 2.6 meaning remission
American College of Rheumatology (ACR) response criteria | Date of inclusion (baseline), day 7, after 6 and 12 weeks
  Change from Baseline in fulfilling the ACR response criteria indicating therapy response rate in percent (none, ACR20, ACR50 or ACR70)
Simplified Disease Activity Index Score (SDAI) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
  Change from Baseline in the SDAI, range from 0 to 86 with assumed range from 0.1 to 10mg/dL for CRP. Higher values mean a higher disease activity and below of 34 meaning remission.
Bio-electrical impedance analysis (BIA) | Date of inclusion (baseline), after 6 and 12 weeks
  Estimation of the body composition via bio-electrical impedance analysis (body fat and visceral fat in %)
Bio-electrical impedance analysis (BIA) | Date of inclusion (baseline), after 6 and 12 weeks
  Estimation of the body composition via bio-electrical impedance analysis (muscle mass in kg)
Abdominal circumference | Date of inclusion (baseline), after 6 and 12 weeks
Resting blood pressure | Date of inclusion (baseline), after 6 and 12 weeks
Pulse rate | Date of inclusion (baseline), after 6 and 12 weeks
Differential blood count | Date of inclusion (baseline), day 7, after 6 and 12 weeks
Hepatic transaminases (GPT, GOT) and Gamma glutamyl transpeptidase (y-GT) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
  * GPT in units per liter (U/L)
  * GOT (U/L)
  * y-GT (U/L)
Total protein in grams per liter (g/L) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
Creatinine in µmol per liter (µmol/L) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
Creatine kinase (U/L) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
Estimated glomerular filtration rate (eGFR) in milliliter per minute (mL/min) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
Electrolytes | Date of inclusion (baseline), day 7, after 6 and 12 weeks
  * calcium in millimol per liter (mmol/L)
  * potassium (mmol/L)
  * sodium (mmol/L)
Erythrocyte sedimentation rate (ESR) in millimeters per hour (mm/h) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
CRP in milligram per liter (mg/L) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
International normalized ratio (INR) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
Partial thromboplastin time (PTT) in seconds (s) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
Lactate dehydrogenase (LDH) (U/L) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
Blood lipids and fasting glucose | Date of inclusion (baseline), day 7, after 6 and 12 weeks
  * triglycerides (mmol/L)
  * total cholesterol (mmol/L)
  * LDL (mmol/L)
  * HDL (mmol/L)
  * fasting glucose (mmol/L)
Uric acid (µmol/L) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
Rheumatoid factor (IgM) | Date of inclusion (baseline)
Anti-cyclic citrullinated peptide (anti-CCP) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
Phenotyping of immune cells | Date of inclusion (baseline), day 7, after 6 and 12 weeks
  Determination of cytometric parameters that indicate changes in cell activation or quantitative changes in the absolute and/or relative size of subpopulations (e.g. classical/intermediate/non-classical monocytes, naïve and memory T-cells, B-cell differentiation to plasmablasts/-cells) Gene expression analysis of immune cells with Affymetrix whole genome microarrays and RNAseq to search for transcriptional patterns and markers that help to identify relevant immune cell (sub-)populations, which are not yet included in the cytometric phenotyping screen
Metabolic plasma metabolites | Date of inclusion (baseline), day 7, after 6 and 12 weeks
  Metabolic plasma metabolites of carbon metabolism with a blood spot extract using metabolomics (GC / MS)
Urine analysis (10 ml midstream urine) | Date of inclusion (baseline), day 7, after 6 and 12 weeks
Gut microbiome | Date of inclusion (baseline), day 7, week 6 and week 12
  Molecular typing of the extremely individual intestinal microbiota composition by sequencing of stool material (16S-, 18S-, ITS-amplicon sequencing, metagenomics, metatranscriptomics) and performing proteomics and metabolomics to characterize fasting and diet induced changes of the so far insufficiently characterized gut microbiota related molecular components in a subgroup of patients
Sociodemographic Measurements | Date of inclusion (baseline)
  age, education level, household income, employment status, marital status, language spoken, complete family history of rheumatoid arthritis in first- and second-degree relatives, current and previous illness and co-morbidities, and current medications
Medication intake | Date of inclusion (baseline), after 6 and 12 weeks
  Systematized documentation of medication, main and secondary diagnoses using CRF
Analgetics intake | Up to 12 weeks
  Systematized documentation of analgetic medication on a daily basis using a diary
Documentation of Behavioral Factors | Up to 12 weeks
  Documentation of digestion, menstruation, compliance on diet and extraordinary events on a daily basis using a diary
Quantification of Behavioral Factors | Up to 12 weeks
  Documentation of occupational stress, domestic stress, interpersonal conflicts on a daily basis using a diary via visual analog scale (VAS), range from 0 to 10 while higher values meaning a higher grade of stress
Quantification of Behavioral Factors | Date of inclusion (baseline), after 6 and 12 weeks
  Nicotine, Alcohol, Physical Inactivity, Coffee and Media Consumption via Likert Scales, range from 0 to 5 while higher values meaning a higher grade of agreement
Food selection | Date of inclusion (baseline), after 4 and 9 weeks
  Nutritional history via dietary record (each for 3 days)
Dietary Behaviour | Date of inclusion (baseline), after 6 and 12 weeks
  Modified FFQ recording dietary behaviour such as mealtimes, frequency of food intake, food preferences, fasting experiences
The Hannover Functional Ability Questionnaire (Funktionsfragebogen Hannover, FFbH-R) | Date of inclusion (baseline), after 6 and 12 weeks, after 6 months
  Change from Baseline in the FFbH-R, range from 0 to 100 % while higher values meaning a higher grade of functional capacity
Mood questionnaire (Profile of Mood States, POMS) | Date of inclusion (baseline), after 6 and 12 weeks, after 6 months
  Change from Baseline in Emotional Distress will be measured using the German Version of the Profile of Mood States (POMS) short version (35 items, 7-point Likert scale; 0=not at all, 6=extremely). It has 65 items and 6 domains: depression [range 0 - 98], vigour-activity [range 0 - 49], fatigue [range 0 - 49], and anger-hostility [range 0 - 49]. The total mood disturbance score is derived by subtracting the vigour-activity score from the the sum of scores from the other subscales. Lower scores indicate more stable mood profiles.
Stress questionnaire (Cohen Perceived Stress Scale, CPSS) | Date of inclusion (baseline), after 6 and 12 weeks, after 6 months
  Change from Baseline in the CPSS, range from 0 to 4 in each item. Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the positively stated items and then summing across all scale items while higher values meaning a higher grade of perceived stress.
Quality of Life questionnaire (WHO-5) | Date of inclusion (baseline), after 6 and 12 weeks, after 6 months
  Change from Baseline in the WHO-5, range from 0 to 100 % while higher values meaning a higher grade of well-being

OTHER OUTCOMES:
Final questionnaire to record tolerability of fasting and nutrition, adverse effects | after 12 weeks
  Measurement of tolerability of fasting and nutrition as well as adverse effects via Likert Scales, range from 0 to 5 while higher values meaning a higher grade of agreement

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charité Hochschulambulanz für Naturheilkunde, Immanuel Krankenhaus Berlin
Locations (2):
- Germany (2):
  - Charité Hochschulambulanz für Naturheilkunde, Immanuel Krankenhaus Berlin, Berlin
  - Charité University, Berlin, Department of Rheumatology and Clinical Immunology, Berlin

IPD SHARING:
Plan to Share IPD: Yes
The study protocol is to be published open access. On publishing the outcomes, the anonymized individual participant data that underlie the reported results, as well as the statistical code, will be made available to scientific investigators who issue a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 10 years after publication of primary results
Access Criteria: * scientific objective (non-commercial)
  * sound methodology

REFERENCES:
- [Derived] Hartmann AM, Dell'Oro M, Spoo M, Fischer JM, Steckhan N, Jeitler M, Haupl T, Kandil FI, Michalsen A, Koppold-Liebscher DA, Kessler CS. To eat or not to eat-an exploratory randomized controlled trial on fasting and plant-based diet in rheumatoid arthritis (NutriFast-Study). Front Nutr. 2022 Nov 2;9:1030380. doi: 10.3389/fnut.2022.1030380. eCollection 2022. PMID 36407522
- [Derived] Hartmann AM, Dell'Oro M, Kessler CS, Schumann D, Steckhan N, Jeitler M, Fischer JM, Spoo M, Kriegel MA, Schneider JG, Haupl T, Kandil FI, Michalsen A, Koppold-Liebscher DA. Efficacy of therapeutic fasting and plant-based diet in patients with rheumatoid arthritis (NutriFast): study protocol for a randomised controlled clinical trial. BMJ Open. 2021 Aug 11;11(8):e047758. doi: 10.1136/bmjopen-2020-047758. PMID 34380725